CLINICAL TRIAL: NCT06515808
Title: Effects of GlideScope, Pentax Airway Scope, and Macintosh Blade on the Incidence of Postoperative Sore Throat: A Cohort Study of 10,382 Patients
Brief Title: Effects of Three Airway Instruments on the Incidence of Postoperative Sore Throat
Status: Completed | Type: Observational
Sponsor: Fu Jen Catholic University Hospital (Other)
Responsible Party: Principal Investigator, Sung, Chao-Hsien, Attending Anesthesiologist, Fu Jen Catholic University Hospital
Other Study IDs: FJUH111171
Record Dates: First submitted 2024-07-14; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Sore-throat
Keywords: Glidescope; Macintosh Blade; Airway Scope; Postoperative sore throat; General Anesthesia
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Direct Laryngoscope Group: Patients receiving tracheal intubation with direct laryngoscope
  Interventions: Device: Direct Laryngoscope
- GlideScope Group: Patients receiving tracheal intubation with GlideScope
- AirwayScope Group: Patients receiving tracheal intubation with AirwayScope

INTERVENTIONS:
Device: Direct Laryngoscope — Patient receiving tracheal intubation with direct laryngoscope, GlideScope or Airway Scope
  Other Names: GlideScope AVL; AirwayScope S100
  Groups: Direct Laryngoscope Group

SUMMARY:
Postoperative sore throat (POST) is a common complaint after general anesthesia. POST is defined by the presence of a self-reported foreign body sensation or a painful sensation in the throat after general anesthesia. This condition may affect recovery and patient satisfaction and is associated with many factors, including intubation tools. Previous studies have reported conflicting results on POST. This retrospective cohort study, with sample size of 10,382 patients, was conducted to confirm the hypothesis that the use of video laryngoscopy (VL) is associated with a lower incidence of POST compared with direct laryngoscopy (DL).

DETAILED DESCRIPTION:
Background: Postoperative sore throat (POST) is a common complaint after general anesthesia. POST is defined by the presence of a self-reported foreign body sensation or a painful sensation in the throat after general anesthesia. This condition may affect recovery and patient satisfaction and is associated with many factors, including intubation tools. Previous studies have reported conflicting results on POST. This retrospective cohort study, with sample size of 10,382 patients, was conducted to confirm the hypothesis that the use of video laryngoscopy (VL) is associated with a lower incidence of POST compared with direct laryngoscopy (DL).

Methods: Data were extracted from a prospectively maintained quality improvement database. A total of 10,382 patients were included in the study. Statistical analysis was conducted for comparisons of demographic characteristics and to determine the effect of intubation tools on the incidence of POST.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving inpatients surgery and general anesthesia with tracheal intubation

Exclusion Criteria:

* Having difficult airway,

  * Anticipated difficult airway:

    1. Abnormal cervical spine movement or temporomandibular joint movement
    2. Airway-compromising masses such as tumors, cysts, or hematomas
    3. A Mallampati score greater than 3
    4. A thyromental distance of less than 6 cm
    5. A lesion below vocal cord
    6. A previously identified difficult airway
  * Unexpected difficult airway

    1. difficult mask ventilation
    2. difficult vocal cord visualization after multiple attempts of laryngoscopy
* Receiving laryngeal surgery, such as laryngeal biopsy, laryngeal microsurgery, laryngoplasty or vocal cord surgery,
* Not being extubated at the end of anesthesia,
* Being pregnant,
* Being under 20 years of age,
* American Society of Anesthesiologists (ASA) physical status class greater than 3.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent inpatient surgeries and general anesthesia with endotracheal tubes, intubated with direct laryngoscope, Pentax AirwayScope or GlideScope, during the period from January 1, 2018, to December 30, 2019, were included for the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 10382 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative sore throat (POST) | 12 to 24 hours after general anesthesia is finished
  POST is defined by the presence of a self-reported foreign body sensation or a painful sensation in the throat after general anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Hsien Sung, MD, Principal Investigator — Fu Jen Catholic University Hospital, Fu Jen Catholic University
Locations (1):
- Fu Jen Catholic University Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are not openly available due to institutional privacy guidelines but may be available from the corresponding author upon written request identifying the requestor, and the purpose and proposed use of the shared data.

REFERENCES:
- [Derived] Fu CH, Sung CH. Effects of GlideScope, Pentax Airway Scope, and Macintosh Blade on the incidence of postoperative sore throat: a cohort study of 9,881 patients. BMC Anesthesiol. 2024 Nov 12;24(1):409. doi: 10.1186/s12871-024-02798-x. PMID 39533185